CLINICAL TRIAL: NCT02867839
Title: A Randomized, Multicentral, Controlled, Phase III Study to Compare Adjuvant Chemotherapy With S-1 Plus Oxaliplatin to S-1 Alone After Curative Distal Gastrectomy in Locally Advanced Gastric Cancer
Brief Title: Adjuvant Chemotherapy With S-1 Plus Oxaliplatin Versus S-1 Alone in Locally Advanced Gastric Cancer
Acronym: RESCUE-GC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The number of patients enrolled was much less than expected
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESCUE-GC-2016
Record Dates: First submitted 2016-08-04; First posted 2016-08-16 (Estimated); Last update posted 2024-12-03 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Adjuvant chemotherapy; S1; Oxaliplatin; Survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: postoperative Oxaliplatin plus S-1 (Experimental): Patients in arm A will receive standard distal gastrectomy with D2 lymphadenectomy first, and 8 cycles of adjuvant Oxaliplatin plus S-1 (SOX) later.
  Oxaliplatin: 130mg/m2, iv drip for 2h, d1, q3W S-1: 40~60mg bid, po, d1~14, q3W (6 months)
  Interventions: Drug: Oxaliplatin plus S-1
- B: postoperative S-1 only (Active Comparator): Patients in arm B will receive standard distal gastrectomy with D2 lymphadenectomy first, and 16 cycles of adjuvant S-1 later.
  S-1: 40~60mg bid, po, d1~14, q3W (12 months)
  Interventions: Drug: S-1 only

INTERVENTIONS:
Drug: Oxaliplatin plus S-1 — 8 cycles of adjuvant chemotherapy with Oxaliplatin plus S-1
  Other Names: SOX
  Arms: A: postoperative Oxaliplatin plus S-1
Drug: S-1 only — 16 cycles of adjuvant chemotherapy with S-1 only
  Other Names: S-1
  Arms: B: postoperative S-1 only

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of S-1 plus Oxaliplatin versus S-1 only as adjuvant chemotherapy after curative distal gastrectomy in patients with locally advanced gastric cancer.

DETAILED DESCRIPTION:
The study is a multi-central, controlled, randomized Phase III trial. The protocol has been approved by the Ethics Committee of Beijing Cancer Hospital. The primary endpoint is the 3-year progression-free survival (PFS) rate. The secondary endpoints are the overall survival (OS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* sign written informed consent form
* age ≥ 18 years, ≤69 years
* ECOG status: 0~2
* pathologically confirmed gastric cancer at stage II or IIIA (AJCC 7th version)
* negative peritoneal cytology
* underwent curative distal gastrectomy with D2 lymph node dissection
* no prior antitumor treatment is allowed, including chemotherapy, radiotherapy, immune therapy or target therapy
* adequate organ function as defined below: Hematologic ANC ≥ 2*109/L, Platelets ≥ 100*109/L, AST and ALT ≤ 2.5×ULN, TBIL ≤ 1.5×ULN.

Exclusion Criteria:

* be enrolled in other clinical trials
* underwent prior antitumor treatment
* allergic reaction to S-1 or oxaliplatin
* abnormal GI tract function
* female in pregnancy or lactation, or refuse to receive Contraception measures during chemotherapy
* other situation to be judged not adaptive to the study by investigators

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
disease-free survival | 5 years

SECONDARY OUTCOMES:
overall survival | up to 5 years
  To evaluate the 1-year, 3-year and 5-year overall survival of GC patients underwent post-operative chemotherapy of S-1 compared with post-operative SOX
Incidence of Treatment-Emergent Adverse Events [Safety] | 1 year
  The incidence of chemotherapy related adverse events in GC patients underwent post-operative chemotherapy of S-1 compared with post-operative SOX

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, MD, Study Chair — Peking University Cancer Hospital & Institute
Locations (15):
- China (15):
  - Cancer Hospital Chinese Acadamy of Medical Sciences, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing General Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Daliang Medical University, Daliang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu X, Chen L, Du Y, Fan B, Bu Z, Wang X, Ye Y, Zhang Z, Xiao G, Li F, He Q, Li G, Shen X, Xiong B, Zhu L, Liu J, Liu L, Wu T, Zhou J, Zhang J, Zhao G, Wang X, Liang P, Wang X, Zhang Y, Wu X, Zhang J, Ji X, Zong X, Fu T, Jia Z, Ji J. Postoperative chemotherapy with S-1 plus oxaliplatin versus S-1 alone in locally advanced gastric cancer (RESCUE-GC study): a protocol for a phase III randomized controlled trial. Chin J Cancer Res. 2017 Apr;29(2):144-148. doi: 10.21147/j.issn.1000-9604.2017.02.07. PMID 28536493